CLINICAL TRIAL: NCT00930995
Title: Angiotensin Receptor Blockade an Anti-Fibrotic Intervention in Patients With Chronic Hepatitis C
Brief Title: Angiotensin Receptor Blockade as an Anti-Fibrotic Intervention in Patients With Chronic Hepatitis C
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not Awarded
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sripriya Balasubramanian MD MPH, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN-05SBala-01-B
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Candesartan
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — 16mg po daily
  Other Names: Atacand
  Arms: A
Drug: Placebo — once daily
  Arms: B

SUMMARY:
Hepatitis C is the most common reason for liver transplantation in the United States and affects nearly 4 million Americans. Treatments for hepatitis C are available but are poorly tolerated and are not always effective. Morbidity and mortality from hepatitis C are related to the development and progression of hepatic fibrosis to cirrhosis and end stage liver disease. Efforts to block progression of liver disease would thus result in prevention of morbidity and mortality as well as costs incurred by the health system in the care of these conditions.

Scar tissue in the liver is secreted by a type of cell, called the stellate cell, in an activated state. This cell carries a receptor for angiotensin, a hormone, when activated. If this receptor is blocked, the cell becomes inactive and does not participate in scar tissue formation. Thus, we hypothesize that using a drug such as candesartan, which blocks angiotensin receptors, should result in less scar tissue formation in the livers of patients with hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 21 and older
* Patients with viral hepatitis C that are not on interferon based therapy.
* Detectable viral load
* Baseline biopsy within six months or willing to undergo biopsy prior to drug initiation
* At least grade 2 inflammation on biopsy, fibrosis of stage 1 or higher
* Willing to undergo biopsy at the end of treatment
* No interferon for at least 6 months prior to or after initial biopsy for study

Exclusion Criteria:

* Renal impairment defined by a serum creatinine of >1.8
* Congestive heart failure
* Hepatocellular cancer
* Concurrent treatment with pentoxyfylline, steroids, interferon alpha or interferon gamma.
* Active psychosis (affective disorders without loss of reality testing acceptable)
* Active IV drug use
* Prior liver transplant
* Pregnancy
* Decompensated cirrhosis as defined by the presence of ascites, hepatic encephalopathy or coagulopathy with an INR>1.4
* HIV seropositivity
* Hypotension defined by a baseline systolic blood pressure of less than 90mm of mercury
* Contraindication to ARB use or allergy to medication
* Treatment with potassium sparing diuretics

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Primary: • Stellate cell activity by alpha SMA stain quantitated by morphometry | 48 weeks
• Hepatic fibrosis by morphometry | 48 weeks

SECONDARY OUTCOMES:
Surrogate markers for fibrosis (liver TGF-beta levels, serum procollagen-III peptide levels) | 48 weeks
Functional status- Albumin, INR, T. Bilirubin, MELD score | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sripriya Subramanian, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente, Roseville, California
  - Kaiser Permanente, Sacramento, California